CLINICAL TRIAL: NCT04887337
Title: Early arthroscoPic Stabilization veRsus rehabilitatiOn of the Shoulder in Adolescents With a trauMatic First-time Anterior Shoulder Dislocation ePisode (PROMPT): A Pilot Randomized Controlled Trial
Brief Title: Early arthroscoPic Stabilization veRsus rehabilitatiOn of the Shoulder in Adolescents With a trauMatic First-time Anterior Shoulder Dislocation ePisode
Acronym: PROMPT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PROMPT
Record Dates: First submitted 2021-05-06; First posted 2021-05-14 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-10

CONDITIONS: Shoulder Dislocation
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arthroscopic stabilization (Active Comparator): Patients will have an initial evaluation with a diagnostic shoulder arthroscopy and examination under anesthesia will be performed to confirm the degree of anterior instability and assess range of motion of the affected shoulder. Diagnostic arthroscopy will commence with the use of 3 standard shoulder portals (posterior viewing and two anterior working portals for suture passing), and a detailed arthroscopic examination will be performed. Once the soft tissue tear (including the labrum, and capsule labrum ligaments) is identified, it will be mobilized using a rasp or elevator and a burr will then be used to create a surface for a bleeding bone bed. Capsulolabral repair will then commence with the labrum fixed to the glenoid using suture anchors (the Bankart repair). Following surgery, subjects in this group will follow the same rehabilitation protocol as the comparison group.
  Interventions: Procedure: Arthroscopic stabilization
- Rehabilitation including a period of immobilization followed by physical therapy (Active Comparator): Subjects in this group will use an internal-rotation shoulder immobilizer, using a standard sling for 6 weeks from the day of enrollment. Subjects will be advised to maintain range of motion (ROM) in the elbow and wrist during this period of time. The immobilizer can be removed for passive pendulum exercises and elbow ROM during the period of immobilization up to 4 times per day. Formal physiotherapy commences at 4 weeks post-enrollment, with a goal of return to activities or sport at 6-months post-enrollment.
  Interventions: Other: Rehabilitation including a period of immobilization followed by physical therapy

INTERVENTIONS:
Procedure: Arthroscopic stabilization — Early arthroscopic stabilization with Bankart repair
  Arms: Arthroscopic stabilization
Other: Rehabilitation including a period of immobilization followed by physical therapy — Rehabilitation including a period of immobilization followed by physical therapy
  Arms: Rehabilitation including a period of immobilization followed by physical therapy

SUMMARY:
Each year within Canada and the US, more than 30,000 children and adolescents will have an injury to their shoulder resulting in a shoulder dislocation. Although the current practice is to manage this initial dislocation without surgery, the vast majority of these children and adolescents will, unfortunately continue to have instability episodes of their shoulder. Recurrent instability can cause damage to the bones and cartilage that form the shoulder resulting in potentially more difficult surgical stabilization, and possibly long-term sequela. To that effect, there is increasing interest to consider early surgical stabilization in this population. This pilot randomized controlled trial (RCT) will evaluate the feasibility of conducting a larger RCT assessing the effect of early arthroscopic stabilization compared to rehabilitation on the rate of repeat shoulder dislocations (recurrent instability), pain, and shoulder function among adolescents (aged 12-18 years) with first-time shoulder dislocations. These patients will be followed for one year.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between the ages of 12 and 18, inclusive
2. Patients with a first-time traumatic anterior glenohumeral dislocation within the past 3 months
3. Anterior glenohumeral dislocation confirmed by radiography, reduction required by medical personnel, or demonstration of anterior apprehension on physical examination following injury to the shoulder
4. MRI or MRA demonstrating disruption of the glenohumeral soft tissues (including the labrum, periosteum, or inferior glenohumeral ligament) relating to instability
5. Patients who have the ability to speak, understand, and read English
6. Provision of informed consent (age 18) or parental consent (ages 12-17, inclusive)
7. Provision of informed child assent (ages 12-17, inclusive)

Exclusion Criteria:

1. Previous dislocation episodes or instability of the affected shoulder
2. Previous surgeries involving the affected shoulder
3. History or clinical exam findings of generalized ligamentous laxity (defined as a Beighton score of 4 or more points)
4. History of multi-directional instability of either shoulder
5. Concomitant fracture of the tuberosity, humerus, or glenoid (excluding a Bankart or Hill Sachs lesion)
6. Bony Bankart lesion exceeding 15% of the glenoid surface (using the best-fit circle method on MRI)
7. Hill Sachs lesion exceeding 15% of the humeral diameter (Measured on transaxial slice of MRI similar to Salomonsson et al.)
8. A neurological injury of the affected arm
9. Patients who will likely have problems, in the judgement of the investigator, with maintaining follow-up
10. Any other reason(s) the investigator feels is relevant for excluding the patient

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2025-10-24 (Actual); Study Completion 2025-10-24 (Actual)

PRIMARY OUTCOMES:
Rate of recurrent shoulder dislocation | 12 months
  Recurrent shoulder dislocations will be defined as an episode of repeat anterior shoulder dislocation either requiring reduction by medical personnel, an x-ray confirming anterior dislocation of the shoulder, or the requirement of surgical management of recurrent instability.

SECONDARY OUTCOMES:
Visual Analogue Scale | 12 months
  100-point pain scale, range 0-100, higher score indicates worse pain.
Pediatric and Adolescent Shoulder and Elbow Survey | 12 months
  The Pediatric and Adolescent Shoulder and Elbow Survey has recently been adopted as a shoulder and elbow function scale designed specifically for children and adolescents aged 10-18, and has shown to be well received and understood in this age group. The total score - 100 maximum points - is weighted 50% for pain and 50% for function.
Euro-Qol 5 Dimensions Youth | 12 months
  The Euro-Qol 5 Dimensions Youth comprises 5 dimensions of health (mobility, self-care [looking after myself], usual activities, pain/discomfort, and anxiety/depression [feeling worried, sad or unhappy]). Score range 0-100, higher score indicating worse outcomes.
Rate of adverse events (other than recurrent shoulder dislocations) | 12 months
  Defined as any symptom, sign, illness, or experience that develops or worsens in severity during the course of this study.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No